CLINICAL TRIAL: NCT05219201
Title: Effectiveness of Partial-body Cryotherapy on the Fatigue of Patients With Multiple Sclerosis During Readaptation Stay
Brief Title: Effectiveness of Cryotherapy on the Fatigue of Patients With Multiple Sclerosis
Acronym: CRYOSEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Collaborators: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-RCB 2021-A02526-35
Record Dates: First submitted 2022-01-07; First posted 2022-02-01 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: cryotherapy; fatigue; quality of life; spasticity; quality of sleep; depression symptoms
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Muscle Spasticity; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham cryotherapy full time patient (inpatient) (Sham Comparator): Patients benefiting from 15 session of "sham" partial-body cryotherapy session (-30°C) during their full-time rehabilitation stay
  Interventions: Device: partial-body cryotherapy chamber session
- sham cryotherapy part-time hospitalized patient (outpatient) (Sham Comparator): Patients benefiting from 15 session of "sham" partial-body cryotherapy session (-30°C) during their part-time rehabilitation stay
  Interventions: Device: partial-body cryotherapy chamber session
- cryotherapy full-time hospitalized patient (inpatient) (Active Comparator): Patients benefiting from 15 session of "sham" partial-body cryotherapy session (-120°C) during their full-time rehabilitation stay
  Interventions: Device: partial-body cryotherapy chamber session
- cryotherapy part-time hospitalized patient (outpatient) (Active Comparator): Patients benefiting from 15 session of "sham" partial-body cryotherapy session (-120°C) during their part-time rehabilitation stay
  Interventions: Device: partial-body cryotherapy chamber session

INTERVENTIONS:
Device: partial-body cryotherapy chamber session — The cryotherapy procedure consisted of a 2-3 min stay in the cryotherapy chamber:
  * at -30°C for sham cryotherapy session
  * at -120°C for cryotherapy intervention session. For Inpatients, cryotherapy session will be performed daily, late in the afternoon, excluding saturdays and sundays, during 3 weeks. (15 sessions) For outpatient, cryotherapy session will occured late in the afternoon each day care (15 sessions).
  Other Names: CRYO00002 ICE X- Cryosauna; local cryotherapy devices DM Class IIb

SUMMARY:
the aim of the study is to evaluate the effectiveness of partial-body cryotherapy (PBC) on the symptoms of patients with multiple sclerosis during a rehabilitation stay.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic heterogeneous disease with an unpredictable clinical course. Symptoms can include paralysis, ataxia, spasticity, incontinence and fatigue syndrome.

Fatigue is considered to be the most prevalent and disabling of the symptoms at all stages of the illness and its occurs in 70-80% of patients. This characteristic of the disease directly impacts the quality of life of patients, affecting their social and physical well being.

Physical rehabilitation is often prescribed in the management of MS, and is recognized to improve modifiable impairments in MS.

However, the benefit of physical activities may be limited by heat stress also named Uhthoff syndrome frequently observed in patients with MS.

Cryotherapy is commonly used as a method to relieve pain and inflammation without marked side effect in respect to contraindication. However well designed studies on PBC in patients with MS are still too sparse.

The investigators propose to evaluate the effectiveness of PBC on the symptoms of MS patients during a rehabilitation stay in out- or inpatients.

ELIGIBILITY:
Inclusion Criteria:

* men and woen over 18 years old and under 65 years old
* with multiple sclerosis
* 0-6 points in the expanded disability states scale (EDSS)
* with MS in remission (at least 6 months since the last relapse)
* able to understand and respect the protocol and its requirement
* who signed the consent prior to any other procedure protocol

Exclusion Criteria:

* major patients under guardianship/curators/legal protection
* pregnant patients
* patients with contraindication for cryotherapy
* patients unable to complete the entire program
* patients with substantial change in pharmacological treatment the month before the start of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Fatigue syndrome | change from baseline (T0) to discharge between 3 to 5 weeks (T1), and 1 month (T2), 3 months (T3) and 1 year (T4) after hospitalization
  evaluation of the fatigue syndrome using the fatigue severity scale score (FSS).
  The scale ranges in value from 9 to 63 with high scores indicating the worse outcome.

SECONDARY OUTCOMES:
spasticity symptom | change from baseline (T0) to discharge between 3 to 5 weeks (T1), and 1 year (T4) after hospitalization
  evaluation of the spasticity syndrome using the Ashworth score The scale ranges in value from 0 to 4 with high scores indicating the worse outcome.
quality of Life evaluation | change from baseline (T0) to discharge between 3 to 5 weeks(T1), and 1 month (T2), 3 months (T3) and 1 year (T4) after hospitalization
  evaluation of the quality of life using the Medical Outcome Study Short Form 36 health survey (MOS-SF36) score.
  The higher score indicating the better outcome.
pain evaluation | change from baseline (T0) to discharge between 3 to 5 weeks(T1), and 1 month (T2), 3 months (T3) and 1 year (T4) after hospitalization
  evaluation of pain syndrome using the visual pain scale The scale ranges in value from 0 to 10 with high scores indicating the worse outcome.
quality of sleep | change from baseline (T0) to discharge between 3 to 5 weeks(T1), after 1 month (T2), 3 months (T3) and 1 year (T4)
  evaluation of sleep quality using the Pittsburgh scale. The scale ranges in value from 0 to 21 with high scores indicating the worse outcome.
depression symptoms | change from baseline (T0) to discharge between 3 to 5 weeks(T1), and 1 month (T2), 3 months (T3) and 1 year (T4) after hospitalization
  evaluation of depression symptoms using the Beck scale. The scale ranges in value from 0 to 39 with high scores indicating the worse outcome.
physician's global assessment-physical endurance | change from baseline (T0) to discharge between 3 to 5 weeks (T1), and 1 year (T4) after hospitalization
  Evaluation of the 6MWT (6 minutes walk test). High scores indicating the better outcome.
habit changes after rehabilitation stay | change from baseline (T0) to 1 month (T2), 3 months (T3) and 1 year (T4) after hospitalization
  Examining habit changes concerning cold therapy after rehabilitation stay using qualitative questionnaire consisting of a small number of direct and meaningful questions (mode and frequency of use).
physician's global assessment-dynamic balance test | change from baseline (T0) to discharge between 3 to 5 weeks (T1), and 1 year (T4) after hospitalization
  Evaluation of the TUG (Time up to go) . High scores indicating the worse outcome.
physician's global assessement-static balance test | change from baseline (T0) to discharge between 3 to 5 weeks (T1), and 1 year (T4) after hospitalization
  Evaluation of the OLS (one leg stance) High scores indicating the better outcome.

OTHER OUTCOMES:
Evaluation of cryotherapy effectiveness on fatigue syndrome in accordance to hospitalisation pattern | change from baseline (T0) to discharge between 3 to 5 weeks (T1)
  Primary outcome will be analyzed separately in outpatient versus inpatient in order to determine whether hospitalisation pattern may impact the effectiveness of cryotherapy on fatigue.
  evaluation of the fatigue syndrome using the fatigue severity scale score (FSS).
  The scale ranges in value from 9 to 63 with high scores indicating the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Bourseul, MD, Principal Investigator — Fondation Ildys
Locations (1):
- Centre de Perharidy, Roscoff, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawik M, Kowalska J, Rymaszewska J. The effectiveness of whole-body cryotherapy and physical exercises on the psychological well-being of patients with multiple sclerosis: A comparative analysis. Adv Clin Exp Med. 2019 Nov;28(11):1477-1483. doi: 10.17219/acem/104529. PMID 30968613
- [Background] Bouzigon R, Grappe F, Ravier G, Dugue B. Whole- and partial-body cryostimulation/cryotherapy: Current technologies and practical applications. J Therm Biol. 2016 Oct;61:67-81. doi: 10.1016/j.jtherbio.2016.08.009. Epub 2016 Aug 27. PMID 27712663
- [Background] Radecka A, Knyszynska A, Luczak J, Lubkowska A. Adaptive changes in muscle activity after cryotherapy treatment: Potential mechanism for improvement the functional state in patients with multiple sclerosis. NeuroRehabilitation. 2021;48(1):119-131. doi: 10.3233/NRE-201535. PMID 33386821
- [Background] Zielinska-Nowak E, Wlodarczyk L, Kostka J, Miller E. New Strategies for Rehabilitation and Pharmacological Treatment of Fatigue Syndrome in Multiple Sclerosis. J Clin Med. 2020 Nov 7;9(11):3592. doi: 10.3390/jcm9113592. PMID 33171768
- [Background] Miller E, Kostka J, Wlodarczyk T, Dugue B. Whole-body cryostimulation (cryotherapy) provides benefits for fatigue and functional status in multiple sclerosis patients. A case-control study. Acta Neurol Scand. 2016 Dec;134(6):420-426. doi: 10.1111/ane.12557. Epub 2016 Jan 18. PMID 26778452